CLINICAL TRIAL: NCT07251036
Title: Serum Chordecone Concentration in Guadeloupean Population: Impact of a Multidisciplinary Support Program on the Reduction of the Contamination Level.
Acronym: ChlorGua
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de la Guadeloupe (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PAP_RIPH2_2022/01
Record Dates: First submitted 2025-11-14; First posted 2025-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-10

CONDITIONS: Chlordecone Level
Keywords: risk factors; pesticides; Guadeloupe; chlordecone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- guadeloupean subject (Other): All subject overs 18 years of age residing in Guadeloupe invited to participate to the program
  Interventions: Other: CHLORGUA

INTERVENTIONS:
Other: CHLORGUA — The target populations will receive an invitation letter with an information notice and a consent form. The referral physician will explain the program and the research project and prescribe a standardized blood sample test.
  Blood samples will be taken in one of the biology laboratories participating in the project. Serum chordecone test will be performed by the Pasteur Institute of Guadeloupe. Blood samples for biological collection will be sent to the Biological Resource Center, Karubiotec™. The result of the chlordécone level will be sent back to each subject with a recommendation note based on the chlordécone level value. Phone contact information for

SUMMARY:
The French West Indies (Guadeloupe, Martinique) are characterized by a major use of pesticides in bananas plantation from the 1950s. These crops used organochlorine insecticides and especially chlordecone (CLD) from 1972 to 1993. The lack of biotic and abiotic degradation of CLD led to persistent soil pollution, contamination of surface and deep waters, of numerous plant and animal, and of the population. The extent and persistence of CLD contamination over time is a major issue for these territories. An internal reference value (0.4μg/l) was recently determined. Although useful for a population approach, it must be used with caution for the interpretation of an individual result. In response to the strong social demand expressed by the population for access to free chlordecone blood tests, a screening program for blood chlordecone test was authorized by the 2019 French Finance Act.

DETAILED DESCRIPTION:
The target populations will receive an invitation letter with an information notice and a consent form. The referral physician will explain the program and the research project and prescribe a standardized blood sample test.

Blood samples will be taken in one of the biology laboratories participating in the project. Serum chordecone test will be performed by the Pasteur Institute of Guadeloupe. Blood samples for biological collection will be sent to the Biological Resource Center, Karubiotec™. The result of the chlordécone level will be sent back to each subject with a recommendation note based on the chlordécone level value. Phone contact information for those who consented to the study will be forwarded to the research assistant for the questionnaire.

ELIGIBILITY:
* All subject overs 18 years of age residing in Guadeloupe invited to participate to the program by the Regional Health Agency or subjects who requested a test from their doctor in the framework of the ministerial measure.
* Subjects who have read the information note and signed the consent to participate in the study
* Subjects with social security coverage

Exclusion Criteria:

* Refusal to participate
* Person not affiliated with a social security scheme
* Person under legal protection (safeguard of justice, guardianship, curatorship, etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3000 (Estimated)
Dates: Start 2022-06-26 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
chlordecone level | between Day0 to Day15
  ug/l
risk factors | between day 15 and day 45 ,
  chlordeconemia survey

SECONDARY OUTCOMES:
chlordecone level | At 9 months after intervention
  ug/l
chlordecone level | At 18 months after intervention
  ug/l
chlordecone level | at delivery for pregnant women
  ug/l
impact of an intervention | between day 15 to day 45, at month 9 and month 18
  chlordeconemia survey

CONTACTS AND LOCATIONS:
Overall Officials: Jacqueline DELOUMEAUX, Doctor, Principal Investigator — CHU de la Guadeloupe
Locations (1):
- Centre Hospitalier Universitaire de la Guadeloupe, Pointe-à-Pitre, Guadeloupe, Guadeloupe